CLINICAL TRIAL: NCT03580395
Title: Efficacy and Safety of Apatinib Added to Docetaxel and Cisplatin Neoadjuvant Therapy for Patients With Breast Cancer: a Randomized, Parallel Controlled Phase II Trial
Brief Title: Apatinib in Neoadjuvant Therapy for Patients With Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Liu Yunjiang, Professor, Director and Vice-president, Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HebeiMUFH
Record Dates: First submitted 2018-05-21; First posted 2018-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: apatinib; neoadjuvant therapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — apatinib; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apatinib+TP (Experimental): TP neoadjuvant chemotherapy (paclitaxel 165mg/m2 day 1, cisplatin 40mg, day 1-3) combined with apatinib (received TP concurrently with apatinib 500mg, day1-21).
  Interventions: Drug: Apatinib; Drug: paclitaxel; Drug: cisplatin
- TP (Sham Comparator): TP neoadjuvant chemotherapy alone (paclitaxel 165mg/m2 day 1, cisplatin 40mg, day 1-3).
  Interventions: Drug: paclitaxel; Drug: cisplatin

INTERVENTIONS:
Drug: Apatinib — 500mg, day1-21,neoadjuvant therapy
  Arms: apatinib+TP
Drug: paclitaxel — paclitaxel 165mg/m2 day 1
Drug: cisplatin — cisplatin 40mg, day 1-3

SUMMARY:
To verify the role of apatinib in neoadjuvant therapy for breast cancer, the investigators designed a prospective, randomized, parallel-controlled phase II/III trial, to investigate the efficacy and safety of apatinib combined with TP (paclitaxel + cisplatin) or TP regimen alone as neoadjuvant therapy for stage II-III breast cancer treatment. 100 cases of eligible patients were diagnosed by core needle biopsy and immunohistochemistry, with the molecular subtypes of triple-negative, HER2+ or Luminal B, evaluated by pathological complete remission (pCR), objective response rate (ORR), adverse events, disease free survival (DFS) and OS, aiming at providing a new way for neoadjuvant therapy in breast cancer and anti-angiogenic treatment of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. breast invasive carcinoma diagnosed by core needle biopsy, without previous treatments for breast cancer;
2. with the molecular subtypes of triple-negative, HER2+ or Luminal B, confirmed by immunohistochemistry;
3. breast cancer within stage IIb-IIIc, planned to receive neoadjuvant therapy;
4. women aged from 18 to 70 years old;
5. required to have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
6. left ventricular ejection fraction (LVEF) greater than 55% without clinical symptoms or signs of heart failure;
7. Adequate bone marrow, with white blood cell ≥4.0×109 /L，neutrophils ≥2.0×109 /L, platelet ≥100×109 /L, hemoglobin ≥ 90 g/L；
8. Serum creatinine ranges from 44 to 133 mol/L;
9. Glutamic pyruvic transaminase and Glutamic-oxalacetic Transaminase ≤2 times to superior limit of normal value;
10. bilirubin ≤ superior limit of normal value;
11. Expected survival ≥ 12 months;
12. pregnancy tests must be negative, and the couples of patients should agree to use effective contraception during treatment and the following one year;
13. approved by the institutional ethnics committee of the Fourth Hospital of Hebei Medical University, with signature to the Informed consent.

Exclusion Criteria:

1. severe systemic infection;
2. being allergic or intolerant to apatinib, paclitaxel, cisplatin;
3. having received any testing drugs, radiotherapy or other chemotherapy drugs within 30 days before being enrolled in this trial;
4. uncontrolled hypertension, severe heart function;
5. researchers believe that participating in the test does not meet the best interests of the patients (e.g. cause adverse health) or may interfere with the evaluation of response.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is pathological complete remission (pCR) | 4 months
  pCR was defined as no histological evidence of invasive tumor cells in the surgical breast specimen and draining nodes. The presence of residual ductal carcinoma-in situ was not included in the pCR category after neoadjuvant treatment.

SECONDARY OUTCOMES:
The second endpoint includes the objective response rate (ORR) | 4 months
  Evaluation of tumor response was performed by independent evaluators who were blinded to the arm assignment consisted of 2 oncologists and 2 pathologists. Tumor response status was defined according to the Response Evaluation Criteria in Solid Tumors Committee (RECIST). Specifically, the complete response (CR) was defined as the disappearance of all the lesions both in breast specimen and draining nodes; The primary endpoint ORR composed of tumor response classifications of CR and partial response (PR).
Adverse events (AE) | 4 months
  Adverse events (AE) were monitored on an ongoing basis and classified according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 3.0. Patients were assessed for toxicities before each administration., and toxicity was graded accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Yunjiang Liu, MD.,PhD, Principal Investigator — Fourth Hospital of Hebei Medical University, Tumor Hospital of Hebei Province
Locations (1):
- Fourth Hospital of Hebei Medical University, Tumor Hospital of Hebei Province, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided